CLINICAL TRIAL: NCT05329740
Title: Assessment of the Efficacy of Glucocorticoids in Improving Post-operative Organ Dysfunction in Patients With Acute Type A Aortic Dissection(GLAD): a Randomized Controlled Trial
Brief Title: Glucocorticoids for Post-operative Patients With Acute Type A Aortic Dissection (The GLAD Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Guowei Tu, Associated professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2022-030R2
Record Dates: First submitted 2022-03-30; First posted 2022-04-15 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Methylprednisolone; Glucocorticoid; Aortic Dissection; Organ Dysfunction
MeSH Terms: conditions — Aortic Dissection | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid group (Experimental)
  Interventions: Drug: Methylprednisolone Injection
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Methylprednisolone Injection — All eligible patients randomised to the glucocorticoid group will receive intravenous Methylprednisolone for 3 days after surgery. The dosage is 2mg/kg/d on post-operative day 1, 1mg/kg/d on post-operative day 2, and 0.5mg/kg/d on post-operative day 3. The daily dosage will be administered with two injections (12h interval).
  Arms: Glucocorticoid group

SUMMARY:
This study is designed to evaluate the effects of glucocorticoid(GC) on improving post-operative organ dysfunction in patients with acute type A aortic dissection(aTAAD). Subjects with confirmed diagnosis of aTAAD undergoing surgical treatment will be enrolled and 1:1 randomly assigned to receive either glucocorticoids or normal treatment. All patients in the glucocorticoids group will be given methylprednisolone intravenously for 3 days after enrollment. The primary endpoint will be the amplitude of variation of Sequential Organ Failure Assessment score on post-operative day 4 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age above 18 years old (including 18 years old), regardless of gender;
* Confirmed type A aortic dissection with computer tomography and received surgical intervention
* Life expectancy > 3 days after surgery

Exclusion Criteria:

* History of cardiac surgery within the past 3 months or possible iatrogenic aortic dissection
* Bacterial or fungal infection in the past 30 days
* Glucocorticoid or any other anti-inflammatory drug usage in the past 14 days
* Allergic to glucocorticoid
* Pregnant
* Implantation of ICD or permanent pacemaker
* Patients diagnosed with malignant tumor undergoing chemotherapy and immunotherapy.
* Patients with pre-operative severe liver dysfunction (CTP grade C)
* Patients with pre-operative renal insufficiency (patients receiving renal replacement therapy before surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Amplitude of variation of SOFA score on post-operative day 4 compared to baseline | Within 4 days on admission to CSICU

SECONDARY OUTCOMES:
In-hospital mortality | Up to 30 days
Duration of ICU stay | Up to 30 days
Duration of mechanical ventilation | Up to 30 days
Duration of hospital stay | Up to 30 days
The proportion of patients receiving RRT | Up to 30 days
  Use of Renal Replacement Therapy(RRT)
The duration of RRT will be compared between two groups. | Up to 30 days
  Use of Renal Replacement Therapy(RRT)
Incidence of Tracheostomy | Up to 30 days
Incidence of Post-operative infection | Up to 30 days
Changes in Inflammation markers | Within 3 days on admission to CSICU
  Inflammation markers include IL-1, IL2R, IL-6 and TNFa
Rate of Composite outcome | Up to 30 days
  In-hospital mortality or Duration of ICU stay longer than 30 days or The need for tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China